CLINICAL TRIAL: NCT02466009
Title: Regorafenib in Adults 70 Years or Older With Metastatic Colorectal Cancer: A Phase II Study
Brief Title: Regorafenib in Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Aram Hezel, Principal Investigator, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 55555
Record Dates: First submitted 2015-04-09; First posted 2015-06-09 (Estimated); Results first posted 2021-04-06 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Colorectal cancer; metastatic colorectal cancer; colorectal adenocarcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Regorafenib (Experimental): 120 mg qd, 3 weeks on/1 week off (each cycle is 28 days)
  Three 40 mg tablets should be taken in the morning with approximately 8 fluid ounces (240 mL) of water after a low-fat (< 30% fat) breakfast.
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Regorafenib — Regorafenib 120 mg (3 tablets) each day for 21 days of a 28 day cycle with the possibility of an increase in the dose to 160 mg (4 tablets).
  Other Names: Stivarga

SUMMARY:
The purpose of the study is to measure high grade (3-5) toxicity of regorafenib and to monitor the impact of treatment with regorafenib on the quality of life in older adults with metastatic colorectal cancer.

DETAILED DESCRIPTION:
Subjects will be asked to participate in the study because they are aged 70 or older and require treatment for colorectal cancer that has spread to other parts of the body and has not gotten better with other treatment. Subjects will undergo some initial tests to ensure that they meet all criteria necessary to participate in the study. Once the subject has completed initial testing and meets eligibility criteria, the subject will begin treatment with 120 mg of regorafenib (3 tablets) each day for 21 days (3 weeks) in a 28 day cycle (4 weeks). After the first cycle, the doctor will discuss the possibility of increasing the dose to 160 mg (4 tablets) each day for 21 days (3 weeks) in a 28 day cycle (4 weeks) based on the subjects health status. During the study, assessments will be performed to monitor the subjects tolerance and response to the treatment. Regorafenib will continue as long as the subject is tolerating the treatment and the subjects colorectal cancer is either responding to treatment or remains stable.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed colorectal adenocarcinoma
* Measurable metastatic disease.
* Age +/> 70
* Progression on standard therapy, not a candidate for further chemotherapy or patient declines other options
* Life expectancy >/= 12 weeks
* Able to understand and willing to sign written informed consent.
* Laboratory requirements:
* Total bili ≤ 1.5 x upper limit or normal
* Alanine aminotransferase & Asparate aminotransferase ≤ 2.5 x upper limit or normal
* Serum creatinine ≤ 1.5 x upper limit or normal
* International normalized ratio/prothrombin time ≤ 1.5 x upper limit or normal
* Platelet count ≥ 100,000, hemoglobin ≥ 9 g/dL
* Absolute neutrophil count ≥ 1,500. Blood transfusion to meet the inclusion criteria not be allowed.
* Glomerular filtration rate ≥ 60 ml/min
* Subjects of childbearing potential must agree to use adequate contraception beginning at the signing informed consent form until at least 3 months after the last dose of study drug.
* Must be able to swallow and retain oral medications

Exclusion Criteria:

* Currently receiving other systemic therapy for metastatic colorectal cancer
* Previous assignment to treatment during this study. Subjects permanently withdrawn from study participation will not be allowed to re-enter study.
* Uncontrolled hypertension despite optimal medical management
* Active or clinically significant cardiac disease.
* Evidence or history of bleeding diathesis or coagulopathy
* Any hemorrhage or bleeding event ≥ grade 3 within 4 weeks.
* Subjects with thrombotic, embolic, venous, or arterial events, such as cerebrovascular accident, deep vein thrombosis or pulmonary embolus within 6 months of informed consent
* History of other active malignancy within past 2 years.
* Patients with phaeochromocytoma
* Known history of human immunodeficiency virus infection or current chronic/active hepatitis B or C infection.
* Ongoing infection > grade 2
* Symptomatic metastatic brain or meningeal tumors
* Presence of non-healing wound, non-healing ulcer, or bone fracture
* Renal failure requiring hemo- or peritoneal dialysis
* Dehydration ≥ grade 1
* Patients with seizure disorder requiring medication
* Persistent proteinuria ≥ grade 3 Interstitial lung disease with ongoing signs and symptoms at the time of informed consent
* Pleural effusion or ascites that causes respiratory compromise, grade 2 dyspnea
* History of organ allograft including corneal transplant
* Known or suspected allergy or hypersensitivity to the study drug
* Any malabsorption condition
* Any condition which makes the subject unsuitable for trial participation
* Substance abuse, medical, psychological, or social conditions that may interfere with the subject's participation in the study.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2022-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aram Hezel, M.D., Principal Investigator — University of Rochester
Locations (4):
- United States (4):
  - Mayo Clinic, Rochester, Minnesota
  - University of Rochester, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Weinberg BA, Hartley ML, Salem ME. Precision Medicine in Metastatic Colorectal Cancer: Relevant Carcinogenic Pathways and Targets-PART 2: Approaches Beyond First-Line Therapy, and Novel Biologic Agents Under Investigation. Oncology (Williston Park). 2017 Jul 15;31(7):573-80. PMID 28712102

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 31 people were screened and 4 failed screening.
Groups:
- Regorafenib: 120 mg qd, 3 weeks on/1 week off (each cycle is 28 days)
  Three 40 mg tablets should be taken in the morning with approximately 8 fluid ounces (240 mL) of water after a low-fat (< 30% fat) breakfast.
  Regorafenib: Regorafenib 120 mg (3 tablets) each day for 21 days of a 28 day cycle with the possibility of an increase in the dose to 160 mg (4 tablets).
Period: Overall Study
Arm/Group | Regorafenib
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Regorafenib
Number analyzed (Participants) | 27
Age, Continuous [Median (Full Range); unit: years] | 74 [65 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 6
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 27
Number of concomitant medications [Median (Full Range); unit: number of concomitant medications] | 13 [5 to 35]

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Experience Grade 3-5 Toxicity as a Measure of Safety and Tolerability.
Time Frame: From the date of study entry until 30 days after the last dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Regorafenib
Number analyzed (Participants) | 27
Participants | 20

2. Secondary Outcome: Percentage of Subjects Who Responded to Study Treatment
Description: Efficacy outcomes will be response rate (RR), disease control rate (DCR), progression-free survival (PFS) and overall survival (OS). A participant's best response will be classified per RECIST (Response evaluation criteria in solid tumors) criteria into complete response (CR), partial response (PR), stable disease (SD) and progressive disease (PD). If a participant's best response was complete response, partial response, or stable disease they were classified as responding to treatment.
Time Frame: From the date of completion of three cycles of treatment until the date of progression of disease as determined by restaging scans up to 2 years.
Measure: Number; unit: percentage of participants
Arm/Group | Regorafenib
Number analyzed (Participants) | 27
percentage of participants | 3.7

3. Secondary Outcome: Mean Difference in Quality of Life as Assessed by the Functional Assessment of Cancer Therapy-Colorectal (FACT-C) Instrument
Description: The FACT-C instrument is an 11 question survey that asks general questions about the participants digestive system. The instrument scores range from 0-44 with higher scores indicating digestive problems.
Time Frame: baseline and week 4
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Regorafenib
Number analyzed (Participants) | 16
score on a scale | -0.82 [-18.33 to 23.33]

4. Other Pre Specified Outcome: Exploratory Outcome Measure: Percentage of Patients Who Had a Correlation Between Adverse Events and Response Rate
Time Frame: week 4
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 years
Description: Grade 3-5 non-serious adverse events were reported.
Arm/Group | Regorafenib
All-Cause Mortality (participants affected / at risk) | 2/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 20/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regorafenib (N=27)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 4
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Confusion (Psychiatric disorders) | 1
Dizziness (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Investigations - Other (Investigations) | 1
Sinus bradycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 10
hypertension (Vascular disorders) | 16
Thromboembolic event (Vascular disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Intestinal stoma site bleeding (Injury, poisoning and procedural complications) | 1
Anemia (Blood and lymphatic system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-12): https://cdn.clinicaltrials.gov/large-docs/09/NCT02466009/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-14): https://cdn.clinicaltrials.gov/large-docs/09/NCT02466009/ICF_001.pdf